CLINICAL TRIAL: NCT02709122
Title: Are EMS Personnel Prepared to Identify and Decompression of Tension Pneumothorax: A Randomized, Crossover Manikin Trial
Brief Title: Are EMS Personnel Prepared to Identify and Decompression of Tension Pneumothorax
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Łukasz Szarpak, Lukasz Szarpak, Medical University of Warsaw
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 02.010.1MR
Record Dates: First submitted 2016-02-22; First posted 2016-03-15 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Tension Pneumothorax
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- With Tension pneumothorax (Experimental): evaluation of the patient with the existing tension pneumothorax during a simulated CPR - breathing
  Interventions: Device: ThoraQuik atraumatic set for pneumothorax decompression
- Without Tension pneumothorax (Experimental): evaluation of the patient without the existing tension pneumothorax during a simulated CPR - breathing
  Interventions: Device: ThoraQuik atraumatic set for pneumothorax decompression

INTERVENTIONS:
Device: ThoraQuik atraumatic set for pneumothorax decompression — pneumothorax decompression in case it is found in accordance with the actually recommendations

SUMMARY:
The study aims to determine the level of knowledge and skills to recognize and decompression of tension pneumothorax

ELIGIBILITY:
Inclusion Criteria:

* give voluntary consent to participate in the study
* maximum 1 year of work experience in medicine
* paramedics, nurses, physicians

Exclusion Criteria:

* not meet the above criteria
* wrist or low back diseases
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
physiological parameter | intraoperative
  study correctness diagnose of pneumothorax by listening to it with a stethoscope and palpation method. The sounds will be issued by the software of manikin. Correct interpretation of the physiological parameters will be recorded in the survey questionnaire

SECONDARY OUTCOMES:
Procedure of Pneumothorax decompression | intraoperative
  Pneumothorax decompression should be in the 2-3 intercostal space at the upper edge of the rib. subject to evaluation will place the introduction of the cannula.
duration of the procedure | intraoperative
  The time starts from the moment of finding of pneumothorax and ends after its proper decompression
Ease-of-use assessed on a visual analog scale | 1 day
  To access subjective opinion about the difficulty of pneumothorax decompression, participants were asked to rate it on a visual analog scale (VAS) with a score from 1 (extremely easy) to 10 (extremely difficult)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Warsaw, Department of Emergency Medicine, Warsaw, Masovia, Poland

IPD SHARING:
Plan to Share IPD: Undecided